CLINICAL TRIAL: NCT03003520
Title: A Phase 2, Open-label, Multicenter Study to Evaluate the Safety and Clinical Activity of Durvalumab in Combination With Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, Prednisone (R-CHOP) or With Lenalidomide Plus R-CHOP (R2-CHOP) in Subjects With Previously Untreated, High-Risk Diffuse Large B-Cell Lymphoma
Brief Title: A Study of Durvalumab in Combination With R-CHOP or Lenalidomide Plus R-CHOP in Previously Untreated High-Risk Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEDI4736-DLBCL-001; 2015-005173-20 (EudraCT Number)
Record Dates: First submitted 2016-12-22; First posted 2016-12-28 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-04

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: Lymphoma; Diffuse-large B-Cell Lymphoma; Durvalumab; Anti-PD-L1 Antibody; MEDI4736; Immune Checkpoint; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone/Prednisolone; Lenalidomide
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma; Dendritic Cell Sarcoma, Interdigitating | interventions — durvalumab; Rituximab; Doxorubicin; Vincristine; Cyclophosphamide; Prednisone; Adrenal Cortex Hormones; Prednisolone; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DUR + R-CHOP (Experimental): On Day 1 of each 21-day cycle, participants received durvalumab 1125 mg intravenously (IV) followed by R-CHOP (IV rituximab 375 mg/m^2, doxorubicin 50 mg/m^2, vincristine 1.4 mg/m^2 (maximum dose of 2.0 mg total), and cyclophosphamide 750 mg/m^2); Participants also were administered daily oral or IV prednisone/prednisolone 100 mg from Day 1 to 5. Induction treatment continued for a total of 6-8 cycles.
  Participants who achieve a complete response or partial response continue with consolidation therapy treatment consisting of durvalumab monotherapy 1500 mg by IV on Day 1 of each 28-day cycle for up to a total of 12 months.
  Interventions: Drug: Durvalumab; Drug: Rituximab; Drug: Doxorubicin; Drug: Vincristine; Drug: Cyclophosphamide; Drug: Prednisone
- DUR + R2-CHOP (Experimental): Participants start the study on durvalumab in combination with R-CHOP (as described in Arm DUR + R-CHOP). Based on their DLBCL Cell-of-Origin subtype (test typically done between cycles 1 and 2), participants with ABC subtype continue the study taking durvalumab in combination with R2-CHOP. On Day 1 of each 21-day cycle, participants received durvalumab 1125 mg intravenously (IV) followed by R-CHOP. Participants were also administered daily oral or IV prednisone/prednisolone 100 mg from Day 1 to 5. In addition, a daily oral lenalidomide 15 mg was administered from Day 1 to 14 of each 21-day cycle. Induction treatment continued for a total of 6-8 cycles.
  Participants who achieve a complete response or partial response continue with consolidation therapy treatment consisting of durvalumab monotherapy 1500 mg by IV on Day 1 of each 28-day cycle for up to a total of 12 months.
  Enrollment into Arm B was discontinued.
  Interventions: Drug: Durvalumab; Drug: Rituximab; Drug: Doxorubicin; Drug: Vincristine; Drug: Cyclophosphamide; Drug: Prednisone; Drug: Lenalidomide

INTERVENTIONS:
Drug: Durvalumab — Durvalumab was supplied in single use vials as a liquid solution containing 500 mg (nominal) of durvalumab at a concentration of 50 mg/mL to be infused by intravenous (IV) injection.
  Day 1 of each treatment cycle (Induction Period and Consolidation Period) started with the administration of IV durvalumab followed by a 2-hour observation period post infusion.
  Other Names: MEDI4736; IMFINZI™; DUR
Drug: Rituximab — Subsequent to durvalumab infusion, rituximab was administered by IV. Rituximab administration could be split over 2 consecutive days according to local clinical practice. Rapid infusion of rituximab was not allowed in this clinical study.
  Other Names: RITUXAN®
Drug: Doxorubicin — A component of the CHOP therapy administered by IV. CHOP therapy was administered following rituximab.
  Other Names: Adriamycin
Drug: Vincristine — A component of the CHOP therapy administered by IV. CHOP therapy was administered following rituximab.
  Other Names: leurocristine; Oncovin
Drug: Cyclophosphamide — A component of the CHOP therapy administered by IV. CHOP therapy was administered following rituximab.
  Other Names: cytophosphane; Cytoxan
Drug: Prednisone — Prednisone was administered as an IV infusion or by mouth (PO) on Day 1, followed by PO administration on Days 2-5 of each cycle.
  Prednisone could be given prior to other drugs of the CHOP therapy. It was administered after lenalidomide dosing in the R2-CHOP treatment arm.
  Other Names: corticosteroid; prednisolone
Drug: Lenalidomide — Lenalidomide was administered orally in capsule form on Days 1-14 of the DUR+R2-CHOP treatment arm only.
  Other Names: Revlimid®
  Arms: DUR + R2-CHOP

SUMMARY:
This Phase 2, two-arm, open-label study is designed to evaluate the safety, clinical activity, and predictive biomarkers of durvalumab in combination with R-CHOP or R2-CHOP, followed by durvalumab consolidation therapy in previously untreated subjects with high-risk diffuse large B-cell lymphoma (DLBCL). Induction treatment with R-CHOP (± lenalidomide) will last for a total of up to 6 to 8 treatment cycles (21 day cycles), and the total time on study treatment, including durvalumab consolidation, will last up to 12 months.

On 05-Sep-2017, the US FDA has issued a Partial Clinical Hold on this study resulting in the discontinuation of enrollment into Arm B (Durvalumab + Lenalidomide + R-CHOP). After the US FDA Partial Clinical Hold, new eligible participants have been enrolled in Arm A (Durvalumab + R-CHOP).

DETAILED DESCRIPTION:
This research study is conducted in participants with previously untreated, high-risk diffuse large B-cell lymphoma (DLBCL). Patients with high-risk DLBCL typically have insufficient therapeutic outcomes. Therefore, the addition of novel agents to the currently used induction therapy (R-CHOP) is a rational approach to improve therapeutic outcomes in this disease setting.

Based on pre-clinical and clinical observations, it is hypothesized that durvalumab will have activity in DLBCL because the PD 1/PD L1 pathway is involved in the pathophysiology of DLBCL. In particular, the addition of durvalumab may augment the anti-tumor activity of R-CHOP against high-risk DLBCL sub-types.

The safety of durvalumab has already been explored. However, as there is limited clinical experience with durvalumab in DLBCL, the study is divided into two stages:

* A Safety Run-in Stage to evaluate the safety of the treatment combinations until at least 10 subjects are included in each of the two treatment arms
* An Expansion Stage to analyze the clinical activity of the treatment combinations

Results posted following Primary Outcome Completion date are based on a database cut-off of August 2, 2018.

ELIGIBILITY:
Inclusion Criteria:

1. CD20+Diffuse Large B-Cell Lymphoma.
2. Ann Arbor stage 3 or 4 or stage 2 with bulky disease
3. High or high-intermediate disease risk.
4. No prior anti-lymphoma treatment.
5. Subject is willing and able to undergo biopsy.
6. Investigator considers R-CHOP immunochemotherapy appropriate.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
8. Adequate hematology laboratory results (absolute neutrophil count ≥ 1.5 * 10^9/L, platelet count ≥ 75 * 10^9/L, hemoglobin ≥ 10.0 g/dL).
9. Adequate biochemistry laboratory results (aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤ 3.0 * upper limit of normal; bilirubin ≤ 2.0 mg/dL; creatinine clearance of ≥ 40 mL/min).
10. Bi-dimensionally measurable disease (> 2.0 cm).
11. Subject is using effective contraception.

Exclusion Criteria:

1. Diagnosis of lymphoma other than Diffuse Large B-Cell Lymphoma.
2. Composite lymphoma or transformed lymphoma.
3. Primary or secondary Central Nervous System involvement by lymphoma.
4. Seropositive or active viral infection with hepatitis B virus, human immunodeficiency virus or hepatitis C virus.
5. History of other malignancies, unless disease-free for ≥ 5 years.
6. Left ventricular ejection fraction < 50%.
7. Peripheral neuropathy ≥ Grade 2.
8. Prior use of lenalidomide, or monoclonal antibodies against CTLA-4, PD-1, or PD-L1.
9. High risk of developing thromboembolic events, who are unwilling to take venous thromboembolism prophylaxis.
10. Active or prior documented autoimmune or inflammatory disorders within the past 3 years.
11. Current or prior use of immunosuppressive medication within 28 days before start of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2022-04-24 (Actual); Study Completion 2022-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (20):
- United States (7):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Parkview Research Center, Fort Wayne, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester Medical Center, Rochester, New York
  - Mid Ohio Oncology Hematology Inc, Columbus, Ohio
  - Swedish Cancer Institute, Seattle, Washington
- Austria (5):
  - Innsbruck Medical University Department of Internal Medicine, Innsbruck
  - Landeskrankenhaus Salzburg, Salzburg
  - Hanusch Krankenhaus, Vienna
  - Local Institution - 101, Vienna
  - Medical University of Vienna Internalmedicine 1, Hematology, Vienna
- Denmark (3):
  - Aarhus Sygehus, Arhus C
  - Rigshospitalet, Kobenhavns Universitet - Centre for Clinical Intervention Research - The Copenhagen, Copenhagen
  - Odense Universitetshospital, Odense C
- Estonia (2):
  - (North Estonia Medical Centre) - Onkoloogia-ja Hematoloogiakliinik, Tallinn
  - Tartu University Hospital, Tartu
- United Kingdom (3):
  - University Hospital Birmingham, Birmingham
  - Royal Marsden Hospital, London
  - Oxford University Hospitals NHS Trust- Churchill Hospital-Oxford Centre for Respiratory Medicine, Oxford

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome

RESULTS

PARTICIPANT FLOW:
Groups:
- DUR + R-CHOP: Participants receive Induction Therapy (21-day cycles): Durvalumab 1125 mg intravenously (IV) on Day 1 of each 21-day cycle in combination with 6 to 8 cycles R-CHOP (IV rituximab, doxorubicin, vincristine and cyclophosphamide on Day 1; daily oral/IV prednisone/prednisolone from Day 1 to 5).
  Participants then receive Consolidation Therapy (28-day cycles): Durvalumab 1500 mg IV on Day 1 of each 28-day cycle for up to a total of 12 months from C1D1 of induction therapy.
- DUR + R2-CHOP: Participants receive Induction Therapy (21-day cycles): Cycle 1 - induction therapy of durvalumab in combination with R-CHOP (as described in DUR + R-CHOP arm). Starting at cycle 2 - Durvalumab 1125 mg IV on Day 1 of each 21-day cycle in combination with 6 to 8 cycles R2-CHOP (IV rituximab, doxorubicin, vincristine and cyclophosphamide on Day 1; daily oral/IV prednisone/prednisolone from Day 1 to 5; daily oral lenalidomide 15 mg from Day 1 to 14) from the cycle following COO determination until end of induction therapy (Cycle 6 or Cycle 8) or starting Cycle 1 if ABC subtype is identified prior to C1D1.
  Participants then receive Consolidation Therapy (28-day cycles): Durvalumab 1500 mg IV on Day 1 of each 28-day cycle for up to a total of 12 months from C1D1 of induction therapy.
Period: Overall Study
Arm/Group | DUR + R-CHOP | DUR + R2-CHOP
Started | 43 | 3
Completed Induction Treatment | 31 | 3
Completed Consolidation Treatment | 14 | 2
Completed | 14 | 2
Not Completed | 29 | 1
Not completed — Adverse Event | 9 | 0
Not completed — Death | 1 | 0
Not completed — Other reasons | 4 | 0
Not completed — Withdrawal by Subject | 6 | 0
Not completed — Progressive disease | 9 | 1

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | DUR + R-CHOP | DUR + R2-CHOP | Total
Number analyzed (Participants) | 43 | 3 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (12.77) | 67.7 (8.62) | 61.5 (12.57)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 23 | 1 | 24
  >=65 years | 20 | 2 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 1 | 18
  Male | 26 | 2 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 43 | 3 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 42 | 3 | 45
  Not Colected or Reported | 0 | 0 | 0
  Other | 1 | 0 | 1
Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants] — ECOG performance status is used by doctors and researchers to assess how a participant's disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. - 0 = Fully Active (most favorable status); - 1 = Restricted activity but ambulatory; - 2 = Ambulatory but unable to carry out work activities; - 3 = Limited Self-Care; - 4 = Completely Disabled, No self-care (least favorable status)
  Participants
    0 = Fully Active | 16 | 2 | 18
    1 = Restricted activity but ambulatory | 19 | 0 | 19
    2 = Ambulatory but unable to work | 8 | 1 | 9
    3 = Limited Self-Care | 0 | 0 | 0
    4 = Completely Disabled, No self-care | 0 | 0 | 0
Ann Arbor Stage at Diagnosis [Count of Participants; unit: Participants] — The criteria for Clinical Stage (Ann Arbor staging) are as below: - I: involvement of a single nodal region. - II: involvement of 2 or more lymph node regions on the same side of the diaphragm. - III: involvement of lymph node regions on both sides of the diaphragm. - IV: disseminated involvement of 1 or more extra-lymphatic sites with or without associated lymph node involvement.
  Participants
    Stage I | 0 | 0 | 0
    Stage II | 0 | 0 | 0
    Stage III | 9 | 2 | 11
    Stage IV | 34 | 1 | 35
Presence of Bulky Disease at Baseline [Count of Participants; unit: Participants] — Bulky disease refers to the size of the tumor. - Yes = tumor diameter >= 7.0 cm. - No = tumor diameter < 7.0 cm.
  Participants
    Yes | 21 | 2 | 23
    No | 22 | 1 | 23
International Prognostic Index (IPSS) Score [Count of Participants; unit: Participants] — The IPI assesses risk of central nervous system disease according to the following scale: - 0-1: Low risk - 2: Low-Intermediate risk - 3: High-Intermediate risk - 4-5: High risk
  Participants
    0-1: Low risk | 0 | 0 | 0
    2: Low-Intermediate risk | 9 | 0 | 9
    3: High-Intermediate risk | 21 | 0 | 21
    4-5: High risk | 9 | 2 | 11
    Missing | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a Complete Response (CR) at the End of Induction Therapy
Description: The primary efficacy analysis evaluated the complete response rate (CRR) at the end of the induction therapy in the efficacy evaluable population in a comparative manner against historical control. The response to treatment was assessed according to the 2014 International Working Group (IWG) Response Criteria for Non-Hodgkin's Lymphoma (NHL) (Cheson, 2014). CR was defined as a complete metabolic response and radiographic evidence showing target nodes/nodal masses regressed to ≤ 1.5 cm in longest diameter, no new lesions, regression of lymph nodes to normal size, absence of splenomegaly, and absence of bone marrow involvement. Clopper-Pearson two-sided 95% confidence interval is reported. Null hypothesis for the primary endpoint was rejected if the lower limit of the confidence interval for the complete response rate at the completion of the induction therapy in the efficacy evaluable population is above 55%.
Time Frame: From first dose of study drug to end of Induction therapy (Day 1 up to Week 26 - maximum duration of Induction Period).
Population: Efficacy Evaluable Population includes participants who completed at least one cycle of their assigned treatment, had a baseline assessment by CT scan and at least one post baseline tumor response assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DUR + R-CHOP | DUR + R2-CHOP
Number analyzed (Participants) | 37 | 3
percentage of participants | 54.1 [36.9 to 70.5] | 66.7 [9.4 to 99.2]

2. Secondary Outcome: Percentage of Participants Who Responded During Induction and Continued Into Consolidation Therapy (Database Cutoff Date: 02-Aug-2018)
Description: The percentage of participants who achieved a partial response (PR) or complete response (CR) at the end of Induction and continued into consolidation period in the efficacy evaluable population in a comparative manner against historical control. The response to treatment was assessed according to the 2014 International Working Group (IWG) Response Criteria for Non-Hodgkin's Lymphoma (NHL) (Cheson, 2014). CR was defined in outcome #1. PR was defined as a partial metabolic response and radiographic evidence showing ≥ 50% decrease in sum of perpendicular diameters (SPD) of up to 6 target measurable nodes and extranodal sites, no new lesions, spleen must have regressed > 50% in length beyond normal, and residual bone marrow involvement improved from baseline. Clopper-Pearson two-sided 95% confidence interval is reported. Null hypothesis was rejected if the lower limit of the confidence interval for the rate of subjects who continue consolidation therapy out of all subjects.
Time Frame: From first dose of study drug to completion of at least one cycle in the Consolidation Period (Day 1 up to Week 52)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DUR + R-CHOP | DUR + R2-CHOP
Number analyzed (Participants) | 37 | 3
percentage of participants | 67.6 [50.2 to 82.0] | 66.7 [9.4 to 99.2]

3. Secondary Outcome: Percentage of Participants Who Achieved a Clinical Response in the Biomarker Subpopulation for Immunohistochemistry (IHC) CD8 T-Cell Density
Description: Data in the analysis include all participants who received durvalumab, irrespective of the study arm in which they enrolled, because the selected biomarkers have been associated with response in other anti-PD1 or anti-PDL1 studies, such as durvalumab. IHC analysis was performed on the baseline tumor biopsy to quantify CD8 T-cell density. Participants with 'high' values, i.e. above the threshold defined as the median value of 774 cells/mm^2 found in commercial DLBCL samples using matched analytical methods, were predicted to be responders to treatment with durvalumab. The definition of a complete response was that used in the primary outcome.
Time Frame: Biomarker biopsies: Days -28 to Day -1. Clinical response: From first dose of study drug to end of Induction therapy (Day 1 up to Week 26 - maximum duration of Induction Period).
Population: The RNA Biomarker Analysis Set included all Efficacy Evaluable participants who have RNA Sequencing analysis performed on a biopsy sample and collected from the participant before treatment on the protocol. Population included participants who received durvalumab. Samples with whole transcriptome data of low quality were excluded from the set.
Measure: Number; unit: percentage of participants
Groups:
- High Group for CD8 Density: Participants had IHC analysis performed on a biopsy sample collected before treatment on this protocol. The result of their CD8 density evaluation was above threshold,defined as the median of 774 cells/mm^2 found in commercial DLBCL samples using matched analytical methods. Participants with values above threshold were predicted to be responders.
- Low Group for CD8 Density: Participants had IHC analysis performed on a biopsy sample collected before treatment on this protocol. The result of their CD8 density evaluation was below threshold,defined as the median of 774 cells/mm^2 found in commercial DLBCL samples using matched analytical methods. Participants with values below threshold were predicted to be non-responders.
Arm/Group | High Group for CD8 Density | Low Group for CD8 Density
Number analyzed (Participants) | 15 | 11
percentage of participants | 67 | 64
Statistical Analysis 1: Comparison: High Group for CD8 Density vs Low Group for CD8 Density; Test type: Superiority; p > 0.99, Fisher Exact — Significance defined as 0.05
Statistical Analysis 2: Comparison: High Group for CD8 Density vs Low Group for CD8 Density; The Area Under the Receiver Operator Characteristic Curve (AUC-ROC) is the estimated parameter. Responders were compared to non-responders by ranking them according to their CD8 density; Test type: Superiority; p = 0.872, Wilcoxon (Mann-Whitney) — Significance defined as 0.05; AUC-ROC = 0.477

4. Secondary Outcome: Percentage of Participants Who Achieved a Clinical Response in the Biomarker Subpopulation for Immunohistochemistry (IHC) Programmed Death Ligand - 1 (PDL1) Total Percentage
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Groups:
- High Group for PDL1 % of Total Cells: Participants had IHC analysis performed on a biopsy sample collected before treatment on this protocol. The result of their PDL1 % of total cell evaluation was above threshold,defined as the median of 13.8% found in commercial DLBCL samples using matched analytical methods. Participants with values above threshold were predicted to be responders.
- Low Group for PDL1 % of Total Cells: Participants had IHC analysis performed on a biopsy sample collected before treatment on this protocol. The result of their PDL1 % of total cell evaluation was below threshold,defined as the median of 13.8% found in commercial DLBCL samples using matched analytical methods. Participants with values below threshold were predicted to be non-responders.
Arm/Group | High Group for PDL1 % of Total Cells | Low Group for PDL1 % of Total Cells
Number analyzed (Participants) | 20 | 5
percentage of participants | 75 | 20
Statistical Analysis 1: Comparison: High Group for PDL1 % of Total Cells vs Low Group for PDL1 % of Total Cells; Test type: Superiority; p = 0.0403, Fisher Exact — Significance defined as 0.05
Statistical Analysis 2: Comparison: High Group for PDL1 % of Total Cells vs Low Group for PDL1 % of Total Cells; The Area Under the Receiver Operator Characteristic Curve (AUC-ROC) is the estimated parameter. Responders were compared to non-responders by ranking them according to their PDL1 % of total cells; Test type: Superiority; p = 0.523, Wilcoxon (Mann-Whitney) — Significance defined as 0.05; AUC-ROC = 0.583

5. Secondary Outcome: Percentage of Participants Who Achieved a Clinical Response in the Biomarker Subpopulation for Immunohistochemistry (IHC) Programmed Death Ligand - 1 (PDL1) Percentage of Tumor Cells
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Groups:
- High Group for PDL1 % of Tumor Cells: Participants had IHC analysis performed on a biopsy sample collected before treatment on this protocol. The result of their PD-1 % of tumor cell evaluation was above threshold,defined as the median of 6.2% found in commercial DLBCL samples using matched analytical methods. Participants with values above threshold were predicted to be responders.
- Low Group for PDL1 % of Tumor Cells: Participants had IHC analysis performed on a biopsy sample collected before treatment on this protocol. The result of their PDL1 % of tumor cell evaluation was below threshold,defined as the median of 6.2% found in commercial DLBCL samples using matched analytical methods. Participants with values below threshold were predicted to be non-responders.
Arm/Group | High Group for PDL1 % of Tumor Cells | Low Group for PDL1 % of Tumor Cells
Number analyzed (Participants) | 11 | 9
percentage of participants | 64 | 56
Statistical Analysis 1: Comparison: High Group for PDL1 % of Tumor Cells vs Low Group for PDL1 % of Tumor Cells; Test type: Superiority; p > 0.99, Fisher Exact — Significance defined as 0.05
Statistical Analysis 2: Comparison: High Group for PDL1 % of Tumor Cells vs Low Group for PDL1 % of Tumor Cells; The Area Under the Receiver Operator Characteristic Curve (AUC-ROC) is the estimated parameter. Responders were compared to non-responders by ranking them according to their PDL1 % of tumor cells; Test type: Superiority; p = 0.557, Wilcoxon (Mann-Whitney) — Significance defined as 0.05; AUC-ROC = 0.583

6. Secondary Outcome: Percentage of Participants Who Achieved a Clinical Response in the Biomarker Subpopulation for the Interferon Gamma Score (IFNG-Score) From Ribonucleic Acid (RNA)-Sequencing Data
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Groups:
- High Group for RNA IFN Gamma Score: Participants had RNA IFN Gamma Score calculated based on a biopsy sample collected before treatment on this protocol. The result of their RNA IFN Gamma Score was above threshold,defined as the median of 3.28 found in commercial DLBCL samples using matched analytical methods. Participants with values above threshold were predicted to be responders.
- Low Group for RNA IFN Gamma Score: Participants had RNA IFN Gamma Score calculated based on a biopsy sample collected before treatment on this protocol. The result of their RNA IFN Gamma Score was below threshold,defined as the median of 3.28 found in commercial DLBCL samples using matched analytical methods. Participants with values below threshold were predicted to be non-responders.
Arm/Group | High Group for RNA IFN Gamma Score | Low Group for RNA IFN Gamma Score
Number analyzed (Participants) | 7 | 20
percentage of participants | 43 | 60
Statistical Analysis 1: Comparison: High Group for RNA IFN Gamma Score vs Low Group for RNA IFN Gamma Score; Test type: Superiority; p = 0.662, Fisher Exact — Significance defined as 0.05
Statistical Analysis 2: Comparison: High Group for RNA IFN Gamma Score vs Low Group for RNA IFN Gamma Score; The Area Under the Receiver Operator Characteristic Curve (AUC-ROC) is the estimated parameter. Responders were compared to non-responders by ranking them according to their IFNG-Score; Test type: Superiority; p = 0.399, Wilcoxon (Mann-Whitney) — Significance defined as 0.05; AUC-ROC = 0.6

7. Secondary Outcome: Participants With Treatment Emergent Adverse Events (TEAE)
Description: An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen during a study. A serious AE is any AE occurring at any dose that: • Results in death; • Is life-threatening; • Requires or prolongs existing inpatient hospitalization; • Results in persistent or significant disability/incapacity; • Is a congenital anomaly/birth defect; • Constitutes an important medical event. The Investigator assessed the relationship of each AE to study drug and graded the severity according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, Version 4.03): - Grade 1 = Mild (no limitation in activity or intervention); - Grade 2 = Moderate (some limitation in activity; no/minimal medical intervention required); - Grade 3 = Severe (marked limitation in activity; medical intervention required, hospitalization possible); - Grade 4 = Life-threatening; - Grade 5 = Death. Relation to IP is determined by the investigator.
Time Frame: From the date of the first dose of study drug to within 90 days after the last dose of durvalumab or 28 days after the last dose of any investigational product (IP) whichever is greater. (Up to approximately 72 weeks)
Population: Safety Population, which consists of all participants who received at least 1 dose of the study medications. Participants were analyzed in the arm of the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | DUR + R-CHOP | DUR + R2-CHOP
Number analyzed (Participants) | 43 | 3
Participants
  >= 1 Treatment-emergent adverse event (TEAE) | 43 | 3
  >=1 TEAE related to durvalumab | 33 | 3
  >=1 TEAE related to R-CHOP | 40 | 3
  >=1 TEAE related to lenalidomide: number analyzed (Participants) | 0 | 3
  >=1 TEAE related to lenalidomide |  | 3
  >=1 TEAE related to durvalumab or any other IP | 41 | 3
  >=1 TEAE severity grade 3-4 | 37 | 3
  >=1 TEAE severity grade 3-4 related to durvalumab | 18 | 1
  >=1 TEAE severity grade 3-4 related to R-CHOP | 27 | 3
  >=1 TEAE severity grade 3-4 related to lenalidomid: number analyzed (Participants) | 0 | 3
  >=1 TEAE severity grade 3-4 related to lenalidomid |  | 2
  >=1 TEAE severity grade 3-4 related to any IP | 31 | 3
  >=1 TEAE severity grade 5 | 3 | 0
  >=1 TEAE severity grade 5 related to any IP | 0 | 0
  >=1 serious TEAE | 23 | 1
  >=1 serious TEAE related to durvalumab | 10 | 1
  >=1 serious TEAE related to R-CHOP | 10 | 1
  >=1 serious TEAE related to lenalidomide: number analyzed (Participants) | 0 | 3
  >=1 serious TEAE related to lenalidomide |  | 1
  >=1 serious TEAE related to any IP | 14 | 1
  >=1 leading to discontinuation of durvalumab | 13 | 0
  >=1 leading to discontinuation of R-CHOP | 4 | 0
  >=1 leading to discontinuation of lenalidomide: number analyzed (Participants) | 0 | 3
  >=1 leading to discontinuation of lenalidomide |  | 0
  >=1 leading to discontinuation of any IP | 13 | 0
  >=1 leading to interruption of durvalumab | 15 | 2
  >=1 leading to interruption of R-CHOP | 12 | 1
  >=1 leading to interruption of lenalidomide: number analyzed (Participants) | 0 | 3
  >=1 leading to interruption of lenalidomide |  | 2
  >=1 leading to interruption of any IP | 18 | 3
  >=1 leading to infusion interruption of durvalumab | 2 | 0
  >=1 leading to dose reduction of vincristine | 4 | 1
  >=1 leading to dose reduction of lenalidomide: number analyzed (Participants) | 0 | 3
  >=1 leading to dose reduction of lenalidomide |  | 1

ADVERSE EVENTS:
Time Frame: AEs and SAEs were assessed from first dose to 90 days after the last dose of durvalumab or 28 days after the last dose of any other IP, whichever is later (up to approximately 72 weeks) and up to 5 years after enrollment (C1D1) of the last participant to receive lenalidomide (up to approximately 5 years). All-Cause Mortality was assessed in participants from their first dose to their study completion (up to approximately 5 years).
Description: Participants treated with lenalidomide during any stage of the study will be continued to be followed for Second Primary Malignancies (SPM) for up to 5 years after enrollment (C1D1) of the last participant to receive lenalidomide as part of their study treatment.
Arm/Group | DUR + R-CHOP | DUR + R2-CHOP
All-Cause Mortality (participants affected / at risk) | 5/43 | 1/3
Serious Adverse Events (participants affected / at risk) | 23/43 | 1/3
Other Adverse Events (participants affected / at risk) | 43/43 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DUR + R-CHOP (N=43) | DUR + R2-CHOP (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 2 | 0
Pyrexia (General disorders) | 3 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 1 | 0
Meningitis bacterial (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Viral diarrhoea (Infections and infestations) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse large B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DUR + R-CHOP (N=43) | DUR + R2-CHOP (N=3)
Anaemia (Blood and lymphatic system disorders) | 7 | 1
Leukopenia (Blood and lymphatic system disorders) | 7 | 1
Neutropenia (Blood and lymphatic system disorders) | 21 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Vision blurred (Eye disorders) | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 0
Constipation (Gastrointestinal disorders) | 9 | 2
Diarrhoea (Gastrointestinal disorders) | 13 | 1
Dry mouth (Gastrointestinal disorders) | 8 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 18 | 2
Stomatitis (Gastrointestinal disorders) | 8 | 2
Vomiting (Gastrointestinal disorders) | 10 | 0
Chills (General disorders) | 4 | 0
Fatigue (General disorders) | 26 | 2
Mucosal inflammation (General disorders) | 4 | 0
Oedema peripheral (General disorders) | 6 | 1
Pyrexia (General disorders) | 9 | 0
Influenza (Infections and infestations) | 3 | 0
Lung infection (Infections and infestations) | 4 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0
Oral candidiasis (Infections and infestations) | 5 | 0
Oral herpes (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 4 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 1
Blood pressure increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 7 | 0
Decreased appetite (Metabolism and nutrition disorders) | 12 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Histiocytic necrotising lymphadenitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 9 | 1
Dysgeusia (Nervous system disorders) | 6 | 0
Headache (Nervous system disorders) | 11 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 23 | 2
Restless legs syndrome (Nervous system disorders) | 2 | 1
Sensory disturbance (Nervous system disorders) | 0 | 1
Taste disorder (Nervous system disorders) | 4 | 0
Depression (Psychiatric disorders) | 3 | 0
Insomnia (Psychiatric disorders) | 11 | 0
Dysuria (Renal and urinary disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0
Rash (Skin and subcutaneous tissue disorders) | 8 | 1
Hot flush (Vascular disorders) | 3 | 0
Hypotension (Vascular disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
After the US FDA Partial Clinical Hold, enrollment of new participants into Arm B was discontinued. If receiving clinical benefit at the discretion of the Investigator, participants could continue treatment in Arm B after being reconsented. Any newly enrolled participant with DLBCL of ABC COO subtype after the US FDA Partial Clinical Hold could continue induction therapy on Arm A after Cycle 1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/20/NCT03003520/Prot_SAP_002.pdf